CLINICAL TRIAL: NCT00180297
Title: Evaluation of the Success Rate and the Clinical Evolution of a Ventricular Lead Implanted in the Septum Versus the Right Ventricular Apex.
Brief Title: Septal - Success Rate and Clinical Outcome of Septal Implant of Ventricular Defibrillation Lead
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Scientific Corporation (Industry)
Collaborators: Guidant Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: Septal 1.1 / 14.04.2005; 2004/12/012
Record Dates: First submitted 2005-09-12; First posted 2005-09-16 (Estimated); Results first posted 2021-07-01 (Actual); Last update posted 2021-10-14 (Actual); Status verified 2012-09

CONDITIONS: Ventricular Tachycardia; Ventricular Fibrillation
MeSH Terms: conditions — Tachycardia, Ventricular; Ventricular Fibrillation

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- Mid septal site location (Experimental): RV lead is placed at mid septum.
  Interventions: Device: Endotak Reliance G
- Apical site location (Active Comparator): RV lead is placed in apical position
  Interventions: Device: Endotak Reliance G

INTERVENTIONS:
Device: Endotak Reliance G — Reliance G is a defibrillation lead to be placed in the right ventricle.

SUMMARY:
The purpose of this study is to determine the safety and efficacy of the implant of a ICD lead of defibrillation in the septum of the right ventricle

DETAILED DESCRIPTION:
The rate of success at implant and the positive clinical outcomes for the patients implanted with a lead of defibrillation at the septal site would make it possible to recommend this site as a "new standard" for implant of the defibrillation lead in the RV for ICD.

ELIGIBILITY:
Inclusion Criteria:

* ICD indication according to current Guidelines

Exclusion Criteria:

* Indication for cardiac resynchronisation therapy, absence of spontaneous ventricular rhythm, pacemaker dependency

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 215 (Actual)
Dates: Start 2005-04; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Mabo, MD, Principal Investigator — Hôpital Pontchaillou, Rennes, France
Locations (18):
- France (18):
  - CH Amiens, Amiens
  - CHU Angers, Angers
  - CH Besancon, Besançon
  - CHU Clermont Ferrand, Clermont-Ferrand
  - CHU Henri Mandor, Créteil
  - CHU Michalon, Grenoble
  - CH St. Joseph, Marseille
  - CHU La Timone, Marseille
  - CHU Montpellier, Montpellier
  - CHU Nantes, Nantes
  - Nouvelle Clinique Nantaise, Nantes
  - CHU Lariboisière, Paris
  - CHU Pitié Salpitrière, Paris
  - HEGP, Paris
  - Hôpital Pontchaillou, Rennes
  - CHU Rouen, Rouen
  - CHU Rangueil, Toulouse
  - CHU Tours, Tours

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Mid Septal Site Location | Apical Site Location
Started | 107 | 108
Completed (Until 5 years follow-up) | 61 | 67
Not Completed | 46 | 41

BASELINE CHARACTERISTICS:
Population: Intention to Treat with the Endotak Reliance G defibrillation lead - population.
Groups:
- Total: Total of all reporting groups
Arm/Group | Mid Septal Site Location | Apical Site Location | Total
Number analyzed (Participants) | 107 | 108 | 215
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.3 (12) | 59.1 (12.7) | 59.7 (12.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 18 | 34
  Male | 91 | 90 | 181

OUTCOME MEASURES:

1. Primary Outcome: Implant Success Rate at Septal Site
Description: Success of implant procedure: 1. implanted at the randomized site; 2. With electric criteria satisfied: pacing threshold < 1.5V, intrinsic amplitude >3 mV, impedance between 450 and 1800 Ω, shock impedance between 29 and 80 Ω and defibrillation at a maximum of 21J.
Time Frame: At implant
Measure: Count of Participants; unit: Participants
Arm/Group | Mid Septal Site Location | Apical Site Location
Number analyzed (Participants) | 107 | 108
Participants | 97 | 99

2. Secondary Outcome: - The Number of "Low Energy" Shocks (at 11 Joules), Efficient in the VT Zone, in the Population Programmed at This Recommended Value.
Time Frame: 3 months, 6 months, 12 months, 36 months, 60 months
Population: The number of participants analyzed per time frame is excluding those participants that have ended the study before the time frame or for whom visit data is missing
Measure: Count of Participants; unit: Participants
Arm/Group | Mid Septal Site Location | Apical Site Location
Number analyzed (Participants) | 91 | 104
Participants
  3 Months | 0 | 3
  6 Months: number analyzed (Participants) | 75 | 84
  6 Months | 1 | 4
  12 Months: number analyzed (Participants) | 82 | 99
  12 Months | 2 | 7
  36 Months: number analyzed (Participants) | 79 | 85
  36 Months | 2 | 11
  60 Months: number analyzed (Participants) | 61 | 67
  60 Months | 4 | 9

3. Secondary Outcome: The Rate of ATP Success Therapy
Description: in VT zone with at least one efficient ATP
Time Frame: 3 months, 6 months, 12 months, 36 months, 60 months
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Mid Septal Site Location | Apical Site Location
Number analyzed (Participants) | 91 | 104
Participants
  3 Months | 6 | 11
  6 Months: number analyzed (Participants) | 75 | 84
  6 Months | 12 | 14
  12 Months: number analyzed (Participants) | 82 | 99
  12 Months | 19 | 19
  36 Months: number analyzed (Participants) | 79 | 85
  36 Months | 23 | 23
  60 Months: number analyzed (Participants) | 61 | 67
  60 Months | 17 | 20

4. Secondary Outcome: Spontaneous Episodes and Therapy Delivery - at Least One Appropriate Treatment
Time Frame: Discharge, 3 Months, 6 Months, 12 Months, 36 Months, 60 Months
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Mid Septal Site Location | Apical Site Location
Number analyzed (Participants) | 107 | 108
Participants
  Discharge | 1 | 2
  3 Months: number analyzed (Participants) | 91 | 104
  3 Months | 8 | 11
  6 Months: number analyzed (Participants) | 75 | 84
  6 Months | 14 | 17
  12 Months: number analyzed (Participants) | 82 | 99
  12 Months | 21 | 22
  36 Months: number analyzed (Participants) | 79 | 85
  36 Months | 23 | 28
  60 Months: number analyzed (Participants) | 61 | 67
  60 Months | 19 | 23

5. Secondary Outcome: Spontaneous Episodes and Therapy Delivery - at Least One Inappropriate Treatment
Time Frame: Discharge, 3 Months, 6 Months, 12 Months, 36 Months, 60 Months
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Mid Septal Site Location | Apical Site Location
Number analyzed (Participants) | 107 | 108
Participants
  Discharge | 0 | 0
  3 Months: number analyzed (Participants) | 91 | 104
  3 Months | 4 | 3
  6 Months: number analyzed (Participants) | 75 | 84
  6 Months | 3 | 4
  12 Months: number analyzed (Participants) | 82 | 99
  12 Months | 9 | 8
  36 Months: number analyzed (Participants) | 79 | 85
  36 Months | 8 | 6
  60 Months: number analyzed (Participants) | 61 | 67
  60 Months | 8 | 5

6. Secondary Outcome: Evolution of Left Ventricular Ejection Fraction
Description: LVEF at 12 months and the change in LVEF at 12 months compared to implant (in %)
Time Frame: 12 Months
Measure: Mean (Standard Deviation); unit: Percentage of LVEF
Arm/Group | Mid Septal Site Location | Apical Site Location
Number analyzed (Participants) | 82 | 99
Percentage of LVEF
  LVEF at 12 Months | 41.96 (13.81) | 40.57 (14.00)
  LVEF (%) Change from Implant | 5.66 (11.96) | 6.16 (11.96)

ADVERSE EVENTS:
Time Frame: 5 years after device implant
Arm/Group | Mid Septal Site Location | Apical Site Location
All-Cause Mortality (participants affected / at risk) | 20/107 | 27/108
Serious Adverse Events (participants affected / at risk) | 35/107 | 34/108
Other Adverse Events (participants affected / at risk) | 17/107 | 17/108
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mid Septal Site Location (N=107) | Apical Site Location (N=108)
Abdominal (Gastrointestinal disorders) | 2 (2) | 0 (0)
Ablation (Cardiac disorders) | 2 (3) | 0 (0)
Atrial Fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
Aneurysm (Vascular disorders) | 0 (0) | 1 (1)
Angina Pectoris (Cardiac disorders) | 0 (0) | 1 (1)
Angioplasty (Cardiac disorders) | 4 (4) | 0 (0)
Aorto Femoro Bypass (Vascular disorders) | 0 (0) | 1 (1)
Arrhythmic Storm (Cardiac disorders) | 5 (7) | 3 (3)
Artheritis (Infections and infestations) | 0 (0) | 1 (1)
Antivitamin K Overdose (Psychiatric disorders) | 0 (0) | 1 (1)
Bladder Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Bleeding (Vascular disorders) | 1 (1) | 0 (0)
Bypass (Cardiac disorders) | 0 (0) | 1 (1)
Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (2)
Cardioversion (Cardiac disorders) | 2 (2) | 3 (3)
Carotid (Vascular disorders) | 0 (0) | 1 (1)
Cholesystectomy (Hepatobiliary disorders) | 1 (1) | 0 (0)
Connection (Product Issues) | 1 (1) | 0 (0)
Cardiac Resynchronization Therapy - Defibrillator (Cardiac disorders) | 1 (1) | 1 (1)
Cardiovascular Accident (CVA) (Vascular disorders) | 0 (0) | 2 (2)
Dental (General disorders) | 1 (1) | 0 (0)
Defibrillation thhreshold (Cardiac disorders) | 1 (1) | 2 (2)
Diabetes (Endocrine disorders) | 0 (0) | 1 (1)
Dislodgement (Product Issues) | 2 (2) | 1 (1)
Drug (Cardiac disorders) | 6 (8) | 5 (5)
Effusion (Cardiac disorders) | 1 (1) | 0 (0)
End of life (Product Issues) | 3 (3) | 4 (4)
Explant Intracardiac defibrillator (Cardiac disorders) | 1 (1) | 0 (0)
Explant System (Cardiac disorders) | 0 (0) | 1 (1)
Eye (Eye disorders) | 0 (0) | 1 (1)
Failure (Product Issues) | 1 (1) | 1 (1)
Ventricular Fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
Gout (Infections and infestations) | 0 (0) | 1 (1)
Heart Transplant (Cardiac disorders) | 4 (4) | 3 (3)
Hematoma/Infection (Infections and infestations) | 2 (4) | 1 (1)
Hematoma/infection at implant (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
heart Failure (Cardiac disorders) | 5 (9) | 13 (16)
Hypoglycemie (Endocrine disorders) | 1 (1) | 0 (0)
Intracardiac Defibrillator Programming (Cardiac disorders) | 1 (1) | 0 (0)
Infection (Infections and infestations) | 2 (2) | 4 (4)
Left Ventricular assistance (Cardiac disorders) | 1 (1) | 0 (0)
Mitral Valve (Cardiac disorders) | 1 (1) | 0 (0)
Neurologic (Nervous system disorders) | 1 (1) | 2 (2)
Orthopedic (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Orthostatic (Cardiac disorders) | 0 (0) | 1 (1)
Other (Investigations) | 1 (1) | 0 (0)
Oversensing (Product Issues) | 0 (0) | 1 (1)
Pain (Cardiac disorders) | 2 (3) | 0 (0)
Peripheral angioplasty (Cardiac disorders) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumopathy (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pocket infection (Infections and infestations) | 1 (1) | 0 (0)
post sternotomy (Surgical and medical procedures) | 0 (0) | 1 (1)
Pre-transplant (Cardiac disorders) | 0 (0) | 3 (3)
premature End of Life (Product Issues) | 3 (3) | 3 (3)
prostate (Reproductive system and breast disorders) | 1 (1) | 1 (1)
Pulmonary (Respiratory, thoracic and mediastinal disorders) | 2 (4) | 0 (0)
renal angioplasty (Renal and urinary disorders) | 0 (0) | 1 (2)
Renal insufficiency (Renal and urinary disorders) | 0 (0) | 1 (1)
reprogramming (Cardiac disorders) | 1 (1) | 0 (0)
Rhumatism (Infections and infestations) | 0 (0) | 1 (1)
scar dehiscence (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Thyroid (Endocrine disorders) | 1 (2) | 0 (0)
(General disorders) | 0 (0) | 1 (1)
urogenital (Renal and urinary disorders) | 0 (0) | 1 (1)
Vagal syndrome (Nervous system disorders) | 1 (1) | 0 (0)
Ventricular Tachycardia (Cardiac disorders) | 1 (1) | 2 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mid Septal Site Location (N=107) | Apical Site Location (N=108)
Atrial Fibrillation (Cardiac disorders) | 1 (1) | 1 (1)
Angor (Cardiac disorders) | 0 (0) | 1 (1)
Atrial Disorder (Cardiac disorders) | 1 (1) | 0 (0)
Crosstalk (Product Issues) | 1 (1) | 0 (0)
diet (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Dysphagy (Gastrointestinal disorders) | 1 (1) | 0 (0)
healing issue (Surgical and medical procedures) | 1 (1) | 0 (0)
Heart Failure (Cardiac disorders) | 0 (0) | 1 (1)
Impedance > 3000 (Product Issues) | 1 (1) | 0 (0)
Implant (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Inappropriate Therapy (Product Issues) | 1 (1) | 2 (4)
Limit algorhythm (Product Issues) | 2 (3) | 4 (4)
Loss Capture (Product Issues) | 1 (1) | 1 (1)
Neurologic (Nervous system disorders) | 0 (0) | 1 (2)
Oversensing (Product Issues) | 0 (0) | 2 (2)
Pain (General disorders) | 0 (0) | 1 (1)
Psychologic (Psychiatric disorders) | 1 (1) | 0 (0)
Rhythm ID (Product Issues) | 0 (0) | 1 (1)
Shock (Cardiac disorders) | 1 (1) | 0 (0)
Site of puncture (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Smart sensing (Product Issues) | 0 (0) | 1 (1)
Sternotomy wires (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Thyroid (Endocrine disorders) | 1 (1) | 0 (0)
Tricuspid insufficiency (Cardiac disorders) | 0 (0) | 1 (1)
Supraventricular Tachycardia (Cardiac disorders) | 1 (1) | 2 (2)
Tumor (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Inappropriate programming (Product Issues) | 4 (5) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No